CLINICAL TRIAL: NCT00919620
Title: Outcome of Stage-specific Early Intervention for Psychosis in Hong Kong: A Randomized Controlled Study
Brief Title: Stage-specific Case Management for Early Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Kwai Chung Hospital (Other); Kowloon Hospital, Hong Kong (Other); Castle Peak Hospital (Other Government); Shatin Hospital (Other); Tai Po Hospital (Other Government); North District Hospital, Hong Kong (Unknown); United Christian Hospital (Other); Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Eric Y.H. Chen, Professor and Head of Department of Psychiatry, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: jcep-rct
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Psychotic Disorders
Keywords: Psychotic disorders; Psychoses
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- case management (4 yrs) (Experimental): 4-year case management and standard care
  Interventions: Behavioral: stage-specific case-management
- case management (2 yrs) and standard care (2 yrs) (Active Comparator): 2-year case management and standard care
  Interventions: Behavioral: stage-specific case-management
- standard care (4 yrs) (No Intervention): standard care for 4 years

INTERVENTIONS:
Behavioral: stage-specific case-management — Stage-specific case-management for psychosis by designated key-workers according to specified protocol
  Arms: case management (2 yrs) and standard care (2 yrs); case management (4 yrs)

SUMMARY:
One of the commonly adopted strategies in improving outcome in psychotic disorders is by focused, specific and intensive intervention in the initial few years of the disorder. However the effects of intervention and the optimal duration of intervention have seldom been examined in randomized studies. This study uses a randomized controlled study design to investigate the effectiveness of stage-specific case-management in improving outcome of first episode psychotic disorders. It also addresses whether two years of case-management is less effective than four years of case-management over a four year period. A total of 360 subjects, who aged 25 above, and diagnosed with first episode psychotic disorders, will be and randomized into 3 groups: (1) standard care alone without case management, (2) two-year case management, (3) four-year case management. All groups will receive usual standard care treatment. This four-year follow-up study will assess symptoms, functioning, quality of life as well as health economics data.

DETAILED DESCRIPTION:
Psychotic disorder is a debilitating illness which imposes substantial impact to the patients, their families, and the society. The provision of early intervention provides a window of opportunity to minimize the social and economic burden incurred by the illness.

Many previous studies of effectiveness of early intervention used the historical control approach and are subjected to cohort effects. For example, change of medication pattern over time could potentially lead to differences in outcome. In addition, few studies provide longer-term outcome data of treatment program beyond two years. The optimal length of intervention has not been determined, and many programmes used 12-24 month intervention mainly based on resources available. It is also important to ask whether favorable effects of early intervention could be sustained over time. Further analyses will be done to assess whether EI effects are more pronounced in particular subgroups including DUP, age, sex and diagnosis.

The proposed study aims to address these issues by using a randomized controlled design to investigate the longer-term (4 year) outcome of patients with first episode psychosis. The study randomizes 360 patients with first episode psychotic disorders into 3 groups: (1) standard care (outpatient based care with inpatient and community care as required); (2) standard care with 2 years of add-on stage specific case-management (individualized care delivered by designated case managers according to specific protocol); and (3) standard care with 4 years of add-on stage specific case management.

The study hypothesis are: (1) both 2 years and 4 years of case management produce better outcomes than standard care alone; (2) 4 years of case management produces better outcome than 2 years of case management.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia, schizoaffective disorder, schizophreniform psychosis, brief psychosis, psychosis nos or delusional disorder
* Cantonese-speaking Chinese
* Ability to understand the nature of the study and sign informed consent
* Capacity to participate in cognitive testing

Exclusion Criteria:

* Organic Brain disorder
* Known history of intellectual disability

Ages: 26 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2009-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Functioning (social and occupational) | baseline, 6-month, 12-month, 24-month, 36-month, 48-month

SECONDARY OUTCOMES:
Psychotic symptoms | baseline, 6-month, 12-month, 24-month, 36-month, 48-month
  Psychotic symptoms will be assessed using the Positive and Negative Syndrome Scale (PANSS)
Psychotic symptoms | baseline, 6-month, 12-month, 24-month, 36-month, 48-month
  Psychotic symptoms will be assessed using Scale for the Assessment of Positive Symptoms (SAPS)
Psychotic symptoms | baseline, 6-month, 12-month, 24-month, 36-month, 48-month
  Psychotic symptoms will be assessed using Scale for the Assessment of Negative Symptoms (SANS).
Depressive symptoms | baseline, 12-month, 24-month, 36-month, 48-month
  Depressive symptoms will be assessed using the Calgary Depression Scale for Schizophrenia (CDSS).
Neurocognitive functioning | baseline, 12-month, 24-month, 36-month, 48-month
  A battery of neurocognitive tests will be conducted, including Handedness, Trail Making, Wisconsin Card Sorting Test, Semantic Verbal Fluency, Logical Verbal Memory, Visual Patterns Test, Letter Number Span, Monotone Counting, and Soft Neurological Signs.
Health economics | baseline, 6-month, 12-month, 24-month, 36-month, 48-month

CONTACTS AND LOCATIONS:
Overall Officials: Eric YH Chen, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Hui CLM, Wong AKH, Ho ECN, Lam BST, Hui PWM, Tao TJ, Chang WC, Chan SKW, Lee EHM, Suen YN, Lam MML, Chiu CPY, Li FWS, Leung KF, McGhee SM, Law CW, Chung DWS, Yeung WS, Yiu MGC, Pang EPF, Tso S, Lui SSY, Hung SF, Lee WK, Yip KC, Kwan KL, Ng RMK, Sham PC, Honer WG, Chen EYH. Effectiveness and optimal duration of early intervention treatment in adult-onset psychosis: a randomized clinical trial. Psychol Med. 2023 Apr;53(6):2339-2351. doi: 10.1017/S0033291721004189. Epub 2022 Feb 11. PMID 35144700
- [Derived] Puntis S, Minichino A, De Crescenzo F, Cipriani A, Lennox B, Harrison R. Specialised early intervention teams for recent-onset psychosis. Cochrane Database Syst Rev. 2020 Nov 2;11(11):CD013288. doi: 10.1002/14651858.CD013288.pub2. PMID 33135811